CLINICAL TRIAL: NCT04635228
Title: Post-market Real-world Collection Data for the Biodesign® Otologic Repair Graft
Brief Title: Biodesign® Otologic Repair Graft
Status: Completed | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 17-08
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Tympanic Membrane Perforation; Eardrum Perforation
Keywords: tympanoplasty; myringoplasty
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Biodesign Otologic Repair Graft — The Biodesign Otologic Repair Graft is intended for use as grafting material for tympanic membrane perforation closure.

SUMMARY:
The post-market follow-up clinical trial of the Cook® Biodesign® Otologic Repair Graft will follow patients up to 3 months post-implantation to determine the percent of patients with complete closure of the tympanic membrane.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires tympanic membrane closure.

Exclusion Criteria:

* Life expectancy < 12 months
* Known sensitivity to porcine material

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any eligible patient
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Percent of closure | 3 months
  Percent of patients with complete closure of the tympanic membrane.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - IU Health, Indianapolis, Indiana
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University Hospitals-Cleveland, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Gloucestershire Royal Hospital, Gloucester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request after final report has been distributed and ending 5 years after final report has been distributed. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.